CLINICAL TRIAL: NCT05928273
Title: Corheart 6 Left Ventricular Assist System Long Term Follow-up Clinical Evaluation Plan
Brief Title: Corheart 6 LVAS LTFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Core Medical Technology CO.,LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COREMED_LVAD
Record Dates: First submitted 2023-03-17; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-03

CONDITIONS: End-stage Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corheart 6 LVAS (Experimental): Corheart 6 Left Ventricular Assist System (Corheart 6 LVAS) to be used on patients with advanced refractory heart failure.
  Interventions: Device: Corheart 6 Left Ventricular Assist System

INTERVENTIONS:
Device: Corheart 6 Left Ventricular Assist System — Implantation of left ventricular assist device for hemodynamic support

SUMMARY:
This study is to evaluate the safety and effectiveness of the Corheart 6 Left Ventricular Assist System (Corheart 6 LVAS) when used for the treatment of advanced refractory heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patient or legal representative has signed Informed Consent Form (ICF)
3. BSA ≥ 1.0 m2
4. Females of child bearing age must agree to use adequate contraception
5. Patients with NYHA Class IV heart failure symptoms who have failed to be reversed by previous standardized oral treatment with anti-heart failure drugs (ACEI, beta-blockers and diuretics)
6. LVEF ≤ 30%,and at least one of the following conditions occurs:

   1. For those whose condition cannot be reversed or can't be removed by using intraaortic balloon pump (IABP), extracorporeal membrane oxygenator (ECMO) orother short-term mechanical circulation assistance;
   2. Rely on continuous intravenous administration of one or more cardioactive drugs or positive inotropic drugs;
   3. Meeting diagnostic criteria of cardiogenic shock: blood pressure < 90/60mmHg; Cardiac discharge index < 2.0; Pulmonary capillary wedge pressure > 18mmHg

Exclusion Criteria:

1. Etiology of HF due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy,pericardial disease, amyloidosis or restrictive cardiomyopathy.
2. Active, uncontrolled infection confirmed by a combination of clinical symptoms and laboratory tests.
3. In the investigator's judgment, there are technical difficulties that lead to an unacceptable hig surgical risk.
4. The patient was intolerant to anticoagulant or antiplatelet therapy or was unable to receive other perioperative and postoperative treatments that the investigator deemed necessary based on the patient's health condition.
5. Patients require biventricular assist device support.
6. Pregnancies.
7. The patient had moderate to severe aortic insufficiency or a history of mechanical aortic valve implantation, but did not agree or could not be corrected by replacement or replacement of biological valve during LVAD implantation.
8. History of visceral organ transplantation.
9. Have uncorrected thrombocytopenia or severe coagulopathy, such as diffuse intravascular coagulation.
10. TBIL (total bilirubin) > 3.0 mg/dL and serum creatinine (SCr) > 3.0 mg/dL within 48 hours before surgery may require dialysis.
11. History of severe chronic obstructive pulmonary disease (COPD) or restrictive lung disease or a diagnosis of primary pulmonary hypertension。
12. Pulmonary embolism and pulmonary artery systolic blood pressure exceeding 60mmHg within 3 weeks prior to enrollment combined with at least one of the following 2 parameters demonstrated that pulmonary vascular resistance did not respond to drug therapy: pulmonary vascular resistance greater than 8 wood units; The transpulmonary differential pressure exceeds 20mmHg.
13. Established and untreated abdominal or thoracic aortic aneurysm > 5cm in diameter.
14. Severe peripheral vascular disease with resting pain or extremity ulceration.
15. Patients with psychiatric disorders/disorders, irreversible cognitive impairment or psychosocial problems are at risk of failing to comply with research protocols and regulations governing the use of implantable LEFT ventricular assist systems or brain death from various causes.
16. Expect to live less than 1 year if you have a malignant tumor or other disease.
17. Patients participate in any other clinical trials that may influence the results of this study.
18. Other circumstances that are unforeseen and determined by the researcher to be unsuitable.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Survival [ Time Frame: 6 months ] | 6 months
  Patients survived with the device for at least 6 months without disabling stroke (disabling stroke disabling stroke defined as a mRS Score > 3 at 60 days after stroke) and without reoperation (replacement or removal) due to device problems.

SECONDARY OUTCOMES:
Quality of Life (EQ-5D-5L) | Baseline, Month 1, Month 3, Month 6
  The EQ-5D-5L is a standardized measure of health status developed by the EuroQol Group. Patients describe their perceived health status using an analog scale with 0 as the worst health the patient can imagine and 100 as the best health (Visual Analog Score). The patients' scores at one, three and six months were compared to their baseline scores and the resulting positive scores indicated improved quality of life.
Functional Status - Six Minute Walk Test (6MWT) | [ Time Frame: Baseline, Month 1, Month 3, Month 6 ]
  The Six Minute Walk Test(6MWT)measures the distance that a patient can walk in a period of 6 minutes.The distance walked is measured in meters. This test measures the patients' functional status. The more meters a patient can walk over baseline indicates improvement in functional status.
New York Heart Association (NYHA) Classification | Baseline, Month 1, Month 3, Month 6
  NYHA classification relates symptoms to every day activities and patients quality of life. Class 1 = no limitations on physical activity Class 2 - slight limitation of physical activity Class 3 - marked limitation of physical activity Class 4 = unable to carry out any physical activity without discomfort
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline, Month 1, Month 3, Month 6
  Scores range from 0 to 100. Higher scores indicate better quality of life and fewer heart failure symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No